CLINICAL TRIAL: NCT02338115
Title: Defining an Exposure Target for Weekly Paclitaxel Infusion in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Principal Investigator, Daniel Hertz, Research Assistant Professor, University of Michigan Rogel Cancer Center
Other Study IDs: UMCC 2014.002
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum at end of first infusion and 24 hours after Whole blood prior to infusion, at end of infusion and 24 hours after, and every 3-4 weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Weekly paclitaxel treatment group: Breast cancer patients initiating paclitaxel 80mg/m2 weekly x 12 weeks for curative treatment will be followed prospectively for collection of samples and longitudinal neuropathy data.
  Interventions: Drug: Paclitaxel 80mg/m2 weekly x 12 weeks

INTERVENTIONS:
Drug: Paclitaxel 80mg/m2 weekly x 12 weeks
  Other Names: Taxol

SUMMARY:
The purpose of this prospective observational study is to understand the relationship between paclitaxel exposure and development of peripheral neuropathy during treatment.

DETAILED DESCRIPTION:
Paclitaxel is a chemotherapeutic agent commonly used in various tumor types. Paclitaxel efficacy and toxicity are "dose-dependent" meaning that increasing the dose increases treatment efficacy and occurrence of toxicity. When used in the weekly 1-hour infusion regimen paclitaxel is commonly associated with treatment-limiting sensory peripheral neuropathy. At the current standard dose of 80 mg/m2 approximately 20-25% of patients experience treatment-limiting neuropathy.

Drug exposure, not dose, determines treatment efficacy and neuropathy development. When treated with standard doses there is substantial variability in drug exposure meaning some patients are receiving less efficacious treatment than optimal. At this time we do not monitor a patient's exposure because the optimal exposure level has not been defined. The purpose of this study is to prospectively enroll patients for systematic collection of exposure and neuropathy data in order to characterize this relationship. Once the relationship between cumulative exposure and neuropathy has been characterized, this model will be used to define an exposure target in future prospective exposure-guided dose-adjustment trials.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of invasive breast cancer
* Systemic treatment with paclitaxel for curative intent (neoadjuvant, adjuvant, or oligometastatic disease per PI discretion)
* 80 mg/m2 1-hour infusions weekly for up to 12 weeks
* Female sex

  ->18 years old
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Any prior or concurrent treatment with neurotoxic chemotherapy including any taxane, vinca alkaloid, platinum, bortezomib, or thalidomide. Note that concurrent biologic treatment with trastuzumab/pertuzumab for HER2+ patients or prior treatment with Adriamycin/cyclophosphamide are not reasons for exclusion.
* Distant metastatic disease
* Concurrent treatment with duloxetine or enrollment on clinical study of neuroprotective agent
* History of allergic reaction to paclitaxel or cremophor EL
* Current signs or symptoms of severe peripheral neuropathy
* Known family history of hereditary peripheral neuropathy or Charcot-Marie-Tooth disease
* Known current pregnancy

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients receiving weekly 1-hour paclitaxel infusions for curative treatment
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Severe neuropathy | During 12 cycles of paclitaxel treatment (12 weeks for most patients but longer for patients who have treatment delays. Expected maximum 16 weeks of treatment)
  Increase in sensory scale of PRO measure of 5 points or more

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L Hertz, PharmD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States